CLINICAL TRIAL: NCT07099742
Title: A Study of Real-World Effectiveness and Safety of Tirzepatide Among Participants With Obesity With or Without Type 2 Diabetes Mellitus (T2DM) in Bangladesh
Brief Title: Effectiveness and Safety of Tirzepatide Among Participants With Obesity With or Without Type 2 Diabetes Mellitus (T2DM)
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Md. Alimur Reza (Industry)
Responsible Party: Sponsor-Investigator, Dr. Md. Alimur Reza, Study Epidemiologist, Beximco Pharmaceuticals Ltd.
Organization: Beximco Pharmaceuticals Ltd. (Industry)
Other Study IDs: Bex-2502004
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Tirzepatide; Obesity; T2DM
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tirzepatide Group: Participants in this group will receive subcutaneous Tirzepatide administered once weekly at a dose determined by standard clinical practice. The dose may be titrated based on patient tolerability and glycemic response.
  Interventions: Drug: Tirzepatide
- Lifestyle Modification Group: Participants in this group will receive standard counselling on lifestyle modifications, including diet and physical activity, as per routine clinical care.
  Interventions: Behavioral: Life Style Modification

INTERVENTIONS:
Drug: Tirzepatide — Exposure
  Groups: Tirzepatide Group
Behavioral: Life Style Modification — Referent group - Lifestyle interventions, exercise, and diet control
  Groups: Lifestyle Modification Group

SUMMARY:
This is a prospective, multicenter, real-world study conducted in Bangladesh to assess the effectiveness and safety of Tirzepatide compared to structured lifestyle interventions, including dietary modifications and exercise, in obese adults with or without Type 2 Diabetes Mellitus (T2DM).

The study aims to determine whether treatment with Tirzepatide results in superior weight reduction outcomes compared to lifestyle-based approaches. Adult participants (≥18 years) with a body mass index (BMI) ≥25 kg/m² and no prior exposure to GLP-1 receptor agonists will be enrolled at the discretion of the treating physician. Eligible participants will receive either once-weekly Tirzepatide or participate in lifestyle intervention programs aligned with standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes, aged ≥18 years.
* Body mass index (BMI) ≥25 kg/m².
* Naïve to glucagon-like peptide-1 receptor agonist (GLP-1 RA) therapy.
* Self-reported stable body weight (change ≤5 kg) over the past 3 months.

Exclusion Criteria:

* Diagnosis of diabetes other than Type 2 Diabetes Mellitus.
* History of chronic or acute pancreatitis.
* Presence of acute medical conditions, including acute hepatitis, myocardial infarction, stroke, heart failure, febrile illness, or acute diarrheal disease.
* Evidence of significant, uncontrolled endocrine disorders (e.g., Cushing's syndrome, thyroid disorders, adrenal insufficiency, congenital adrenal hyperplasia).
* History or presence of malignancy.
* Active gallbladder disease.
* Female participants who are pregnant, breastfeeding, planning pregnancy, or of childbearing potential, not using adequate contraceptive methods.
* Prior or planned surgical treatment for obesity.
* Use of weight-loss products (including prescription medications, over-the-counter drugs, or herbal preparations) within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult males and females aged 18 years and older who are clinically diagnosed with obesity, with or without Type 2 Diabetes Mellitus. Eligible participants are those who have been prescribed Tirzepatide (2.5 mg, 5 mg, or 7.5 mg) administered subcutaneously once weekly, or who are undergoing structured lifestyle interventions involving extensive exercise and dietary control. Only patients meeting all inclusion criteria and none of the exclusion criteria will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 364 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight at Week 24 in both treatment groups. | Baseline to 24 Weeks
  The percentage change in body weight (kg) from baseline to Week 24 will be assessed and compared between participants treated with Tirzepatide and those undergoing structured lifestyle interventions..
Percentage of participants withdrawn from the study due to adverse events by Week 24 | Up to Week 24
  The proportion of participants in each treatment group (Tirzepatide vs. lifestyle intervention) who discontinue study participation due to adverse events (AEs) will be assessed and compared.

SECONDARY OUTCOMES:
Absolute change in body weight at Week 24 across both treatment groups | Baseline to 24 weeks
  The absolute difference in body weight (kg) from baseline to Week 24 will be assessed and compared between participants treated with Tirzepatide and those undergoing structured lifestyle interventions..
Change from baseline in Body Mass Index (BMI) and waist circumference at Week 24 across both treatment groups | Baseline to Week 24
  The mean change in Body Mass Index (BMI, kg/m²) and waist circumference (cm) from baseline to Week 24 will be evaluated and compared between participants receiving Tirzepatide and those undergoing structured lifestyle interventions.
Percentage of participants achieving ≥15% reduction in body weight from baseline to Week 24 | Baseline to Week 24
  The proportion of participants in each treatment group (Tirzepatide vs. lifestyle intervention) who achieve a ≥15% reduction in body weight from baseline to Week 24 will be assessed and compared
Percent change from baseline in Hemoglobin A1c (HbA1c) at Week 24 | Baseline to Week 24
  The mean percent change in HbA1c from baseline to Week 24 will be evaluated and compared between the Tirzepatide group and the lifestyle intervention group.
Percentage of diabetic participants achieving HbA1c <7% at Week 24 | Week 24
  Among participants with Type 2 Diabetes Mellitus, the proportion achieving an HbA1c level below 7.0% at Week 24 will be assessed and compared between both treatment arms.
Percentage of participants achieving the highest dose of Tirzepatide by Week 24 | Up to Week 24
  The proportion of participants in the Tirzepatide group who are titrated to and maintained on the highest protocol-defined dose (e.g., 7.5 mg) by Week 24 will be evaluated and reported.
Frequency of adverse events (AEs) and serious adverse events (SAEs) reported by Week 24 | Up to Week 24
  The total number of AEs and SAEs reported in each treatment group will be documented and compared over the 24-week period to assess the overall safety profile.
Number of hypoglycemic events reported by Week 24 | Up to Week 24
  The total number of hypoglycemic episodes, as reported by participants or identified through clinical evaluation, will be recorded and compared between both groups.
Number of self-reported gastrointestinal (GI) adverse events by Week 24 | Up to Week 24
  The frequency of self-reported GI-related adverse events (e.g., nausea, vomiting, diarrhea) will be captured through participant diaries or structured interviews and compared across both treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Indrajit Prasad, MBBS, MD(Endo), Principal Investigator — Dhaka Medical College Hospital, Dhaka
Locations (3):
- Bangladesh (3):
  - Trauma Centre, Cumilla., Comilla
  - Dhaka Medical College Hospital, Dhaka, Dhaka
  - Rajshahi Medical College Hospital, Rajshahi, Rajshahi

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared with other researchers due to institutional and regulatory restrictions related to patient confidentiality, data protection regulations, and the absence of a pre-approved data-sharing framework. Additionally, the study is designed as a real-world investigation without predefined provisions for external IPD access. Any future sharing of data will require separate ethical approval and patient re-consent, which are not within the current study's scope.

REFERENCES:
- [Background] Sustaining security's effectiveness as a hospital continues to expand. Hosp Secur Saf Manage. 1996 Sep;17(5):1-3. No abstract available. PMID 10161731
- [Background] Forzano I, Varzideh F, Avvisato R, Jankauskas SS, Mone P, Santulli G. Tirzepatide: A Systematic Update. Int J Mol Sci. 2022 Nov 23;23(23):14631. doi: 10.3390/ijms232314631. PMID 36498958
- [Background] Wadden TA, Chao AM, Machineni S, Kushner R, Ard J, Srivastava G, Halpern B, Zhang S, Chen J, Bunck MC, Ahmad NN, Forrester T. Tirzepatide after intensive lifestyle intervention in adults with overweight or obesity: the SURMOUNT-3 phase 3 trial. Nat Med. 2023 Nov;29(11):2909-2918. doi: 10.1038/s41591-023-02597-w. Epub 2023 Oct 15. PMID 37840095
- [Background] Jastreboff AM, Aronne LJ, Ahmad NN, Wharton S, Connery L, Alves B, Kiyosue A, Zhang S, Liu B, Bunck MC, Stefanski A; SURMOUNT-1 Investigators. Tirzepatide Once Weekly for the Treatment of Obesity. N Engl J Med. 2022 Jul 21;387(3):205-216. doi: 10.1056/NEJMoa2206038. Epub 2022 Jun 4. PMID 35658024
- See also: World Health Organization. Obesity and overweight. Geneva: WHO; 2024. Available from: https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight — https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- See also: World Obesity Federation. World Obesity Day Atlases | Obesity Atlas 2025. London: Global Obesity Observatory; 2025 [cited 2025 Mar 4]. Available from: https://data.worldobesity.org/publications/?cat=23 — https://data.worldobesity.org/publications/?cat=23
- See also: Global Nutrition Report. Bangladesh Nutrition Profile. Bristol: Development Initiatives; 2020. Available from: https://globalnutritionreport.org/resources/nutrition-profiles/asia/southern-asia/bangladesh/ — https://globalnutritionreport.org/resources/nutrition-profiles/asia/southern-asia/bangladesh/
- See also: World Obesity Day. Obesity and NCDs. 2025. Available from: https://www.worldobesityday.org/obesity-and-ncds — https://www.worldobesityday.org/obesity-and-ncds
- See also: World Health Organization. Diabetes. Geneva: WHO; 2024. Available from: https://www.who.int/news-room/fact-sheets/detail/diabetes — https://www.who.int/news-room/fact-sheets/detail/diabetes
- See also: International Diabetes Federation. IDF Diabetes Atlas: Bangladesh [Internet]. Brussels: IDF; 2024. Available from: https://diabetesatlas.org/data-by-location/country/bangladesh/ — https://diabetesatlas.org/data-by-location/country/bangladesh/